CLINICAL TRIAL: NCT04774029
Title: Basivertebral Nerve Block Performed in Conjunction With Vertebral Augmentation for Anesthesia
Brief Title: Basivertebral Nerve Block During Vertebral Augmentation: An Alternative Approach to Intraprocedural Pain Management
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MTH18-017
Record Dates: First submitted 2021-02-17; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Vertebral Compression; Vertebra Compression Fracture; Vertebral Fracture
Keywords: Basivertebral nerve block; Vertebral augmentation; BVN block; Kyphoplasty; nerve block; compression fracture
MeSH Terms: conditions — Spinal Fractures; Fractures, Compression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BVN Block (Experimental): Patients will receive temporary basivertebral nerve block using lidocaine during the vertebral augmentation procedure for osteoporotic compression fracture.
  Interventions: Procedure: Basivertebral nerve block; Drug: Lidocaine induced basivertebral nerve block

INTERVENTIONS:
Procedure: Basivertebral nerve block — Temporary intraosseous basivertebral nerve block using lidocaine
  Other Names: BVN block during vertebral augmentation
Drug: Lidocaine induced basivertebral nerve block — Intraosseous lidocaine basivertebral nerve block
  Other Names: Lidocaine BVN block

SUMMARY:
The goal of this study is to assess the efficacy of lidocaine basivertebral nerve block as intraprocedural anesthesia during vertebral augmentation procedures.

DETAILED DESCRIPTION:
Vertebral compression fractures secondary to osteoporosis can be treated with vertebral augmentation. Since intraprocedural pain is common during vertebral body endplate manipulation, these procedures are often carried out using conscious sedation or general anesthesia. Research has shown that the vertebral endplates are innervated by the basivertebral nerve, which has been successfully targeted via radiofrequency ablation to treat chronic vertebrogenic lower back pain. With this physiology in mind, the investigators will attempt to treated participants with vertebral compression using lidocaine-induced intraosseous basivertebral nerve block as the primary intraprocedural analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Age >50 years old
* Patient must have a diagnosis of osteoporosis on dual energy x-ray absorptiometry (DEXA),
* Patient must have an acute or subacute single level vertebral compression fracture between T10 - L3 as confirmed via magnetic resonance imaging (MRI) or nuclear medicine bone scan,
* Patient must have an initial pain score of greater than or equal to five using a standard 0-10 Visual Analog Scale subjective pain score upon initial consultation.

Exclusion Criteria:

* Pathologic compression fracture, such as due to metastatic disease
* Age >90 years old or <50 years old
* Pregnancy
* Diagnosed Anxiety Disorder
* Diagnosed Depression Disorder
* Diagnosed Psychotic Disorder
* Diagnosed Mental Disease Disorder
* Diagnosed Parkinson's disease/other movement disorders/or cerebellar dysfunction
* Eastern Cooperative Oncology Group (ECOG) score at baseline prior to compression fracture >1
* Back Pain scores at time of initial consult <5, using a standard Visual Analog Scale
* Illicit drug dependence or abuse
* Alcohol dependence or abuse

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Pre-procedure Pain Score | At pre-procedure consultation.
  Subjective pain as measured using a standard Visual Analog Scale (VAS) of 0-10, where 0 represents no pain, and 10 indicates the worst pain of the patient's life. VAS pain scores will be obtained upon preprocedural consultation.
Immediate Post-procedure Pain Score | In the immediate post-procedure period in recover.
  Subjective pain as measured using a standard Visual Analog Scale (VAS) of 0-10, where 0 represents no pain, and 10 indicates the worst pain of the patient's life. VAS pain scores will be obtained immediately post-procedure.
One-week Post-procedure Pain Score | At one-week post procedure follow-up.
  Subjective pain as measured using a standard Visual Analog Scale (VAS) of 0-10, where 0 represents no pain, and 10 indicates the worst pain of the patient's life. VAS pain scores will be obtained at one-week post-procedure follow-up in clinic.
Immediate Post-procedure Satisfaction Score | Assessed at one-week post procedure follow-up.
  Patients will be asked to rate their satisfaction using a subjective Likert scale of 1 - 4, in the immediate post-procedure period during recovery. Satisfaction ratings were defined as follows: 1 = completely dissatisfied, 2 = dissatisfied, 3 = satisfied, 4 = very satisfied.
One-week Post-procedure Satisfaction Score | At one-week post-procedure follow-up.
  Patients will be asked to rate their satisfaction using a subjective Likert scale of 1 - 4, at one week clinical follow-up. Satisfaction ratings were defined as follows: 1 = completely dissatisfied, 2 = dissatisfied, 3 = satisfied, 4 = very satisfied.

SECONDARY OUTCOMES:
Heart rate disturbance | Intraprocedural
  >20% change from baseline heart rate as measured in beats per minute (BPM)
Blood pressure disturbance | Intraprocedural
  >20% change from baseline systolic or diastolic blood pressure as measured in mm of Mercury (mmHg)
Need for additional anesthesia or sedation | Intraprocedural
  Intraprocedural monitoring for patient pain in real time during the procedure. Need for additional pain or sedative medication such as Fentanyl or Versed, at the discretion of the interventional radiologist performing the procedure.
Intraprocedural pain during balloon augmentation | Intraprocedural
  Special attention to patient pain will be assessed during intraprocedural balloon augmentation, as this is often the most painful part of the procedure. Subjective pain as measured using a standard Visual Analog Scale (VAS) of 0-10, where 0 represents no pain, and 10 indicates the worst pain of the patient's life. Additional routine monitoring of pain will take place during the procedure as carried out by the circulating nurse and by the interventional radiologist performing the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Kenny Lien, MD, Principal Investigator — Northwell Health - Mather Hospital
Locations (1):
- Northwell Health Mather Hospital, Port Jefferson, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will be made available upon request at the discretion of the primary investigator.